CLINICAL TRIAL: NCT07138729
Title: Research on the Application of 99mTc-TCR-FAPI SPECT Imaging in Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luo Yaping (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor-Investigator, Luo Yaping, Medical Doctor (M.D.), Chief Physician, Professor, Assistant Director, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI-RA; Categoty C, UBJ10707 (Other: PekingUMCH Talent Cultivation Program)
Record Dates: First submitted 2025-05-07; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid arthritis; 68Ga-FAPI PET / CT; 99mTc-CTR-FAPI SPECT
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPI PET/CT& 99mTc-CTR-FAPI SPECT (Experimental): All enrolled patients will undergo one 99mTc-CTR-FAPI SPECT scan and one 68Ga-FAPI PET/CT scan within a 1-week interval.
  Interventions: Diagnostic Test: 68Ga-FAPI PET/CT and 99mTc-CTR-FAPI SPECT

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI PET/CT and 99mTc-CTR-FAPI SPECT — For 68Ga-FAPI PET/CT scan，each patient was injected with 1.8-2.2 MBq/kg (0.05-0.06 mCi/kg) body weight of 68Ga-FAPI. PET/CT from skull to feet was performed 60±5 min post-injection.
  For 99mTc-CTR-FAPI SPECT scan:each patient was injected with 10-20mCi 99mTc-CTR-FAPI . Planar SPECT scan and SPECT/CT were performed 60±5 min post-injection.

SUMMARY:
This study proposes to evaluate 99mTc-CTR-FAPI SPECT imaging as a cost-effective, low-radiation, and widely accessible alternative to 68Ga-FAPI PET/CT for assessing synovial lesions in RA patients, aiming to validate its diagnostic consistency with both PET/CT and physical examinations while correlating imaging findings with clinical disease activity metrics to establish a practical tool for long-term RA monitoring.

DETAILED DESCRIPTION:
This study will enroll 20 rheumatoid arthritis patients meeting the 2010 ACR/EULAR classification criteria with moderate-to-high disease activity, with all participants undergoing both 99mTc-CTR-FAPI SPECT and 68Ga-FAPI PET/CT imaging for head-to-head comparison.The imaging results of both 99mTc-CTR-FAPI SPECT and 68Ga-FAPI PET/CT were independently interpreted by two nuclear medicine physicians with ≥10 years of diagnostic experience. A joint-by-joint comparison was performed between: (1) FAPI-positive joints identified by 99mTc-CTR-FAPI SPECT versus 68Ga-FAPI PET/CT, and (2) imaging-detected joints versus tender/swollen joints confirmed by physical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. Meet the classification criteria for rheumatoid arthritis of the American College of Rheumatology/European Union for Rheumatology in 2010;
3. The highest disease activity in clinical practice (CDAI or SDAI score

Exclusion Criteria:

1. Patients with other autoimmune diseases;
2. Patients with concurrent tumors;
3. Women who are pregnant or planning to become pregnant, women in the preconception period, pregnant and lactating women, and women with child-rearing plans during the study period; Subjects of childbearing age need to take effective contraceptive measures during the research process;
4. Active infection
5. Suffering from claustrophobia or other mental disorders, with poor compliance resulting in inability to cooperate with this researcher; (6) Situations where other researchers consider it inappropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
The number of affected joints detected by 99mTC-TCR-FAPI SPECT | through study completion, an average of 1 year
  Consistency in detecting affected joints between 99mTc-CTR-FAPI SPECT and 68Ga-FAPI PET/CT interpreted by two nuclear medicine physicians with 10 years of diagnostic experience. The joints that were positive for RA detected by 99mTc-CTR-FAPI SPECT and 68Ga-FAPI PET/CT were compared one by one, and then compared with the joints with tenderness and swelling determined by physical examination.

SECONDARY OUTCOMES:
The correlation of 99mTc-CTR-FAPI SPECT with clinical characteristics | through study completion, an average of 1 year
  (1) Agreement among 99mTc-CTR-FAPI SPECT, 68Ga-FAPI PET/CT, and physical examination in joint assessment; (2) Correlation between imaging findings and clinical disease activity indices.

CONTACTS AND LOCATIONS:
Overall Officials: Yaping LUO, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No